CLINICAL TRIAL: NCT04535219
Title: Effect of Total Sleep Deprivation on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201901937
Record Dates: First submitted 2020-08-24; First posted 2020-09-01 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Participants will have vascular function assessed following total sleep deprivation
  Interventions: Other: Supervised Total Sleep Deprivation
- Group B (No Intervention): Participants will have vascular function assessed following a full night of sleep
- Group C (Experimental): Participants will have vascular function assessed following total sleep deprivation preceded by exercise
  Interventions: Other: Exercise; Other: Supervised Total Sleep Deprivation
- Group D (No Intervention): Participants will have vascular function assessed following a full night of sleep

INTERVENTIONS:
Other: Exercise — 60 minutes of moderate-intensity treadmill exercise (70% of maximal heart rate determined from the maximal graded exercise test)
  Arms: Group C
Other: Supervised Total Sleep Deprivation — Laboratory-monitored total sleep deprivation
  Arms: Group A; Group C

SUMMARY:
Insufficient sleep is associated with an increased risk for cardiovascular disease. The causal mechanisms are currently unknown, but may include endothelial dysfunction. The purpose of this study is to examine the influence of sex and aging on the effects of total sleep deprivation on vascular function and whether exercise training attenuates these effects.

ELIGIBILITY:
Inclusion criteria:

* Males and females
* 20 to 30 and 50 to 60 years of age
* Females will be eumenorrheic at enrollment or postmenopausal for at least 1 year
* No major clinical disease (e.g., diabetes, cardiovascular, liver or chronic kidney disease) to minimize confounding of vascular measures
* Participants will be sedentary (≤3x per week of ≤30 minutes of aerobic exercise/session) or trained (≥5x per week of moderate/vigorous aerobic exercise training)

Exclusion criteria:

* Age <20 or 31 to 49 or >60 years
* Body mass index ≥30 kg/m^2 because obesity may affect vascular function
* Use of medication that may affect vascular measures
* Hormone replacement therapy or hormonal contraceptives within past year
* Use of tobacco products (chewing tobacco, traditional or e-cigarettes) because they may influence vascular function
* Being perimenopausal, pregnant or lactating because may influence vascular function
* Being a shift worker because habitual sleep deprivation and altered circadian rhythm may influence vascular function.
* Not having an "intermediate" chronotype based on the Morningness-Eveningness Questionnaire (MEQ; score <31 or >69) because this would influence the effect of overnight sleep deprivation on vascular function.
* Sleep complaints based on the Pittsburgh Sleep Quality Index (PSQI; score >5) because this would influence the effect of overnight sleep deprivation on vascular function.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-11 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Endothelial function | through study completion, an average of 1 month
  Endothelial function will be determined using brachial artery flow-mediated dilation via high resolution duplex ultrasonography. Reactive hyperemia will be produced by inflating a forearm cuff to ~250 mmHg for 5 minutes followed by rapid deflation.
Microvascular function | through study completion, an average of 1 month
  Microvascular function will be assessed using the forearm blood flow response to submaximal handgrip exercise. Brachial artery blood flow and diameter will be assessed using Doppler ultrasound.

SECONDARY OUTCOMES:
Central arterial stiffness | through study completion, an average of 1 month
  The SphygmoCor XCEL device will be used to measure carotid to femoral pulse wave velocity.
Central arterial hemodynamics | through study completion, an average of 1 month
  The SphygmoCor XCEL device will be used to obtain central pulse wave analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Demetra Christou, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No